CLINICAL TRIAL: NCT02153918
Title: A Phase II Study of Neoadjuvant rFowlpox-PSA (L155)-TRICOM (Prostvac-F/TRICOM) in Combination With rVaccinia-PSA (L155)-TRICOM (Prostvac-V/TRICOM) in Men With Prostate Cancer Undergoing Treatment With Radical Prostatectomy
Brief Title: Vaccine Plus Booster Shots in Men With Prostate Cancer Undergoing Treatment With Radical Prostatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Peter Pinto, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140112; 14-C-0112
Record Dates: First submitted 2014-05-31; First posted 2014-06-03 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: Prostate Cancer; Prostatic Neoplasms; Neoplasms, Prostate
Keywords: Surgery; Neoadjuvant; CD8 Cell Infiltrate Response; CD4 Cell Infiltrate Response; Vaccine
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vaccine Plus Booster Shots (Experimental): PROSTVAC-V/TRICOM followed by PROSTVAC-F/ TRICOM boost monthly until radical prostatectomy or off therapy PROSTVAC
  Interventions: Biological: PROSTVAC-V/TRICOM; Biological: PROSTVAC-F/TRICOM

INTERVENTIONS:
Biological: PROSTVAC-V/TRICOM — A recombinant vaccinia virus vector vaccine containing the genes for human prostatic specific antigen (PSA) and three co-stimulatory molecules.
Biological: PROSTVAC-F/TRICOM — A recombinant fowlpox virus vector vaccine containing the genes for human PSA and three co-stimulatory molecules.

SUMMARY:
Background:

- Some men with prostate cancer have their prostate glands removed. The cancer can still come back. Researchers want to know if receiving a vaccine before prostate removal surgery can lead to less recurrence.

Objective:

- To see if a vaccine and booster shots given to men with prostate cancer before surgery changes the immune cells in the prostate gland.

Eligibility:

- Men age 18 and older who have prostate cancer that has not spread, and who want to have their prostate glands removed as treatment.

Design:

* Participants will be screened by their regular cancer care. They may have a small piece of prostate removed.
* Participants must practice effective birth control before and during the study treatment and for 1 month after the last vaccine booster.
* Participants will have a medical history, physical exam, and blood and liver tests. They will be asked about how they perform daily activities.
* Participants will have a magnetic resonance imaging (MRI) scan of the prostate. The scanner is a metal cylinder in a strong magnetic field. Participants will lie on a table that slides in and out of the scanner.
* Participants will be injected with the vaccine, most likely in the leg. They will be injected with the vaccine booster 3 times over several weeks.
* At each booster visit, participants will have a medical history, physical exam, and blood and liver tests.
* Participants will have another MRI. Then they will have surgery to remove their prostate.
* Participants will have 2 follow-up visits during the year after surgery. They will have a medical history, physical exam, and blood test.

DETAILED DESCRIPTION:
Background

* Adenocarcinoma of the prostate is the most common cancer diagnosis in American males and follows lung cancer as the leading cause of cancer death.
* Vaccine strategies represent a novel therapeutic approach in the treatment for prostate cancer. One potential target for a prostate cancer vaccine is prostatic specific antigen (PSA), due to its restricted expression on prostate cancer and normal prostatic epithelial cells.
* A neoadjuvant approach may be of potential benefit providing prolonged protection via the patient s immune system against future recurrence.
* PROSTVAC is a vaccine that induces strong immune responses, has shown promising evidence of activity in a randomized phase II study (8.5 month improvement in median overall survival) and is currently in phase III clinical testing.
* This vaccine has been tested in locally recurrent prostate cancer with substantial inflammatory infiltrates within the prostate seen following subcutaneous and intraprostatic injection.

Objectives

-The primary objective is to evaluate the post vaccine immunologic cluster of differentiation 4 (CD4) and cluster of differentiation 8 (CD8) cell infiltrate response of a neoadjuvant vaccine strategy in prostatectomy specimens in patients who plan to undergo radical prostatectomy.

Eligibility

* Patients must have biopsy proven prostate cancer and are surgical candidates for radical prostatectomy
* Must be of sufficient good health to be surgical candidates for radical prostatectomy and have elected radical prostatectomy for management of their prostate cancer
* Granulocyte count is greater than or equal to 1,500/mm(3), Platelet is greater than or equal to 50,000/mm(3), hemoglobin (Hgb) is greater than or equal to 8 g/dL, Bilirubin < 1.5mg/dL, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5x upper limit of normal (ULN), Creatinine is less than or equal to 1.5 X ULN
* Pre-intervention biopsy tissue must be available either from outside institution or repeat biopsy

Design

* This study will utilize rV-PSA(L155)-TRICOM (PROSTVAC-V) as a priming vaccination followed by monthly boosting with rF-PSA (L155)-TRICOM (PROSTVAC-F) for 3 months.
* Patients will undergo radical prostatectomy after 4 months of treatment with PROSTVAC-V/F.
* The maximum accrual to the trial will be 27 patients.

ELIGIBILITY:
-INCLUSION CRITERIA

1. Patients must have histopathological documentation of adenocarcinoma of the prostate prior to starting this study and evaluable biopsy tissue (e.g., unstained slides or blocks) available for analysis. If evaluable tissue is not available, the patient must agree to undergo a pre-vaccination prostate biopsy on study as an alternative to having available tissue available.
2. Patients must be a surgical candidate for radical prostatectomy based on standard workup of prostatic specific antigen (PSA), biopsy results, and if necessary supplemental imaging.
3. Patients must have chosen radical prostatectomy as their definitive treatment of choice for management of their prostate cancer.
4. Patients must have a performance status of 0 to 1 according to the Eastern Cooperative Oncology Group (ECOG) criteria
5. No systemic steroid or steroid eye drop use within 2 weeks prior to initiation of experimental therapy. Limited doses of systemic steroids to prevent intravenous (IV) contrast, allergic reaction or anaphylaxis (in patients who have known contrast allergies) are allowed.
6. Hematological eligibility parameters (within one month of starting therapy):

   * Granulocyte count greater than or equal to 1,500/mm(3)
   * Platelet count greater than or equal to 50,000/mm(3)
   * Hemoglobin (Hgb) greater than or equal to 8 g/dL
7. Biochemical eligibility parameters (within one month of starting therapy):

   1. Hepatic function: Bilirubin < 1.5 mg/dl (OR in patients with Gilbert's syndrome, a total bilirubin less than or equal to 3.0 mg/dL), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 times upper limit of normal.-. Creatinine less than or equal to 1.5 X ULN
   2. Creatinine less than or equal to 1.5 X ULN
   3. Patients must be test negative for human immunodeficiency virus (HIV), Hepatitis B and C.
8. Patients must not have other active invasive malignancies within the past 2 years (with the exception of non-melanoma skin cancers) or life threatening illnesses.
9. Patients must be willing to travel to the study site for follow-up visits.
10. Patients must be greater or equal to18 years of age.
11. All patients who have received prior vaccination with vaccinia virus (for smallpox immunization) must not have a history of allergy to the vaccine.
12. Patients must understand and sign informed consent that explains the neoplastic nature of their disease, the procedures to be followed, the experimental nature of the treatment, alternative treatments, potential risks and toxicities, and the voluntary nature of participation.
13. The effects of the study agents used in this protocol on the developing human fetus are unknown. For this reason men must agree to use adequate contraception (abstinence,vasectomy, or female partner use of intrauterine device (IUD), hormonal [birth control pills, injections, or implants], tubal ligation) prior to study entry and for up to one month after the last vaccination.

EXCLUSION CRITERIA

1. Prior splenectomy.
2. The recombinant vaccinia vaccine should not be administered if the following apply to either recipients or, for at least 3 weeks after vaccination, their close household contacts (Close household contacts are those who share housing or have close physical contact):

   * Persons with active or a history of eczema or other eczematoid skin disorders
   * Those with other acute, chronic or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, severe acne or other open rashes or wounds) until condition resolves
   * Pregnant or nursing women; children under 3 years of age
   * Patients should have no evidence, as listed below, of being immunocompromised:
   * HIV positivity due to the potential for decreased tolerance and risk for severe side effects.
   * Hepatitis B or C positivity.
   * Concurrent use of topical steroids (including steroid eye drops) or systemic steroids. This is to avoid immunosuppression which may lead to potential complications with vaccinia (priming vaccination). Nasal or inhaled steroid use is permitted.
3. Patients with known allergy to eggs.
4. Other serious intercurrent illness.
5. Patients with a history of unstable or newly diagnosed angina pectoris, recent myocardial infarction (within 6 months of enrollment) or New York Heart Association class II-IV congestive heart failure.
6. Patients with significant autoimmune disease that is active or potentially life threatening if activated.
7. Patients with clinically significant cardiomyopathy requiring treatment.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-05-31 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2018-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Pinto, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DiPaola RS, Plante M, Kaufman H, Petrylak DP, Israeli R, Lattime E, Manson K, Schuetz T. A phase I trial of pox PSA vaccines (PROSTVAC-VF) with B7-1, ICAM-1, and LFA-3 co-stimulatory molecules (TRICOM) in patients with prostate cancer. J Transl Med. 2006 Jan 3;4:1. doi: 10.1186/1479-5876-4-1. PMID 16390546
- [Background] Gulley JL, Heery CR, Madan RA, Walter BA, Merino MJ, Dahut WL, Tsang KY, Schlom J, Pinto PA. Phase I study of intraprostatic vaccine administration in men with locally recurrent or progressive prostate cancer. Cancer Immunol Immunother. 2013 Sep;62(9):1521-31. doi: 10.1007/s00262-013-1448-0. Epub 2013 Jul 9. PMID 23836412
- [Background] Kantoff PW, Schuetz TJ, Blumenstein BA, Glode LM, Bilhartz DL, Wyand M, Manson K, Panicali DL, Laus R, Schlom J, Dahut WL, Arlen PM, Gulley JL, Godfrey WR. Overall survival analysis of a phase II randomized controlled trial of a Poxviral-based PSA-targeted immunotherapy in metastatic castration-resistant prostate cancer. J Clin Oncol. 2010 Mar 1;28(7):1099-105. doi: 10.1200/JCO.2009.25.0597. Epub 2010 Jan 25. PMID 20100959
- [Derived] Abdul Sater H, Marte JL, Donahue RN, Walter-Rodriguez B, Heery CR, Steinberg SM, Cordes LM, Chun G, Karzai F, Bilusic M, Harmon SA, Turkbey IB, Choyke PL, Schlom J, Dahut WL, Madan RA, Pinto PA, Gulley JL. Neoadjuvant PROSTVAC prior to radical prostatectomy enhances T-cell infiltration into the tumor immune microenvironment in men with prostate cancer. J Immunother Cancer. 2020 Mar;8(1):e000655. doi: 10.1136/jitc-2020-000655. PMID 32269146
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0112.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vaccine Plus Booster Shots
Started | 27
Completed | 26
Not Completed | 1
Not completed — Refused further treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vaccine Plus Booster Shots
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.24 (6.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3
  White | 23
  Mexican, Puerto Rican, Central or So. Amer. or Oth | 2
  Not meeting definition for Hispanic or Latino | 25
  Multi-racial | 1
Region of Enrollment [Number; unit: participants]
  United States | 27
Baseline Prostatic Specific Antigen (PSA) [Mean (Standard Deviation); unit: ng/ml] — PSA levels of 4.0 ng/ml and lower are considered normal.
  ng/ml | 9.66 (10.45)
Magnetic Resonance Imaging (MRI) Prostate Volume at Baseline [Mean (Standard Deviation); unit: cc] — Population: One subject did not have baseline MRI performed.
  cc
    number analyzed (Participants) | 26
    (all) | 45.70 (17.24)
Number of Lesions on MRI at Baseline [Mean (Standard Deviation); unit: lesions] — Population: One patient did not have baseline MRI performed.
  lesions
    number analyzed (Participants) | 26
    (all) | 2.04 (1.21)
Largest Lesion Size at Baseline [Mean (Standard Deviation); unit: cm] — Population: One patient did not have baseline MRI performed.
  cm
    number analyzed (Participants) | 26
    (all) | 1.55 (0.92)
Number of Participants with Gleason Score 6-10 at Baseline [Count of Participants; unit: Participants] — The higher the number on the Gleason scale, the worse the expected outcome.
  Participants
    Gleason score 6-7 (3+4) | 11
    Gleason score 7 (4+3) | 8
    Gleason score 8-10 | 8

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline to After Surgery of Cluster of Differentiation 4 (CD4) and Cluster of Differentiation 8 (CD8) Cell Infiltrates
Description: Immunologic CD4 and CD8 cell infiltrate response of a neoadjuvant prime/boost vaccine strategy in prostatectomy specimens. Prostate biopsy specimens are collected and stained for CD4 and CD8 cells. Quantification is reported as the number of stained cells per micron squared of surface area. Change will be noted by utilizing computer automated staining analysis. Density of cell infiltrate will be calculated and the pre and post vaccine values will be compared to determine response to vaccine.
Time Frame: Baseline (pre vaccination) and approximately week 10
Population: Only 26 participants had available tissue for analysis.
Measure: Median (Inter-Quartile Range); unit: Cell/mm(2)
Arm/Group | Vaccine Plus Booster Shots
Number analyzed (Participants) | 26
Cell/mm(2)
  Median CD4 at baseline | 132.2 [5.856 to 735.2]
  Median CD4 at week 10 | 153.7 [33.71 to 1368]
  Median CD8 at baseline | 105.1 [28 to 637]
  Median CD8 at week 10 | 140.5 [9.45 to 514]

2. Secondary Outcome: Count of Participants With Change in Peripheral Prostatic Specific Antigen (PSA)-Specific T Cell Responses
Description: Change in peripheral prostatic specific antigen (PSA)-specific T cells will be assessed by the enzyme-linked immunospot (ELISPOT) assay. A change of >250 cluster of differentiation 4 (CD4) or cluster of differentiation 8 (CD8) cells producing cytokine or positive for cluster of differentiation 107a (CD107a) in response to PSA post vaccination relative to baseline will be considered evidence of an immunologic response to the vaccine. The number of subjects developing positive PSA-Specific T cell responses with vaccination will be reported.
Time Frame: Baseline (pre vaccination) and week 10
Population: 25/27 pts analyzed because 2x10(6) viable cells are required to setup the stimulation assay for each antigen at each time point and one patient had no viable cells after thawing blood. One patient could not be analyzed due to an experimental error which was a clog in the flow cytometry that occurred during acquisition for the final assay readout.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Plus Booster Shots
Number analyzed (Participants) | 25
Participants
  CD4 CD107a | 4
  CD4 interferon gamma (IFNq) | 2
  CD4 interleukin-2 (IL2) | 1
  CD4 tumor necrosis factor (TNF) | 0
  CD8 CD107a | 0
  CD8 IFNq | 0
  CD8 IL2 | 0
  CD8 TNF | 1

3. Secondary Outcome: Intraprostatic Treg Cell Infiltration With Cluster of Differentiation 4 (CD4)+Forkhead Box P3 (FOX-P3) Staining
Description: Prostate biopsy samples collected at baseline and at surgery after last dose of vaccine will be stained for analysis of immune cell infiltrate. Quantification will be reported as number of stained cells per micron squared of surface area.
Time Frame: Baseline (pre vaccination) and post surgery after last dose of vaccine, approximately week 10
Population: Only 26 subjects had available tissue for analysis.
Measure: Mean (Standard Deviation); unit: Cell/mm(2)
Arm/Group | Vaccine Plus Booster Shots
Number analyzed (Participants) | 26
Cell/mm(2)
  CD4 at baseline | 199.8 (195.3)
  CD4 at surgery after last dose of vaccine | 237.6 (289.9)
  FOX-P3 at baseline | 16.93 (29.3)
  FOX-P3 at surgery after last dose of vaccine | 5.466 (4.524)

4. Secondary Outcome: Prostatic Specific Antigen (PSA) Changes Secondary to Vaccination
Description: A change in PSA secondary to vaccination is defined as an increase or decrease in PSA value beyond the baseline level. PSA levels of 4.0 ng/ml and lower are considered normal.
Time Frame: Baseline (pre vaccination) and approximately week 10
Population: One subject came off-study prior to radical prostatectomy.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vaccine Plus Booster Shots
Number analyzed (Participants) | 26
ng/mL
  PSA at Baseline | 8.94 (9.96)
  PSA at 10 Weeks | 10.18 (15.45)

5. Secondary Outcome: Magnetic Resonance Imaging (MRI) Changes Secondary to Vaccination
Description: MRI of the prostate was performed for changes in imaging characteristics of prostate cancer pre and post vaccination. MRI changes secondary to vaccination is defined as increase or decrease in the size of lesions from baseline (pre-vaccine) measurements.
Time Frame: Baseline (pre vaccination) and approximately week 10
Population: 3 subjects did not have week 10 MRI performed.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Vaccine Plus Booster Shots
Number analyzed (Participants) | 24
cm
  Largest lesion measurement at baseline | 1.58 (0.91)
  Largest lesion measurement at 10 weeks | 1.57 (0.94)

6. Secondary Outcome: Count of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 33 months and 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Plus Booster Shots
Number analyzed (Participants) | 27
Participants | 27

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 33 months and 5 days.
Arm/Group | Vaccine Plus Booster Shots
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 1/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine Plus Booster Shots (N=27)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine Plus Booster Shots (N=27)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 9 (11)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Blurred vision (Eye disorders) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Cholesterol high (Investigations) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (3)
Dysgeusia (Nervous system disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Eye disorders - Other, Blepharitis (Eye disorders) | 1 (1)
Eye disorders - Other, Subconjunctival hemorrhage (Eye disorders) | 2 (2)
Eye pain (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 14 (20)
Fever (General disorders) | 8 (9)
Flu like symptoms (General disorders) | 17 (29)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, H. Pylori (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 1 (1)
Hemoglobin increased (Investigations) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Hypertension (Vascular disorders) | 8 (15)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (4)
Injection site reaction (General disorders) | 27 (83)
Insomnia (Psychiatric disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (4)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — muscle cramps, bilateral lower extremities
Musculoskeletal and connective tissue disorder - Other, muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 5 (7)
Pain in extremity (General disorders) | 4 (4)
Paresthesia (Nervous system disorders) | 5 (5)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Renal and urinary disorders - Other, weak urine stream (Renal and urinary disorders) | 1 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) — subcutaneous air in chest and neck
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) — chest fullness
Sinus bradycardia (Cardiac disorders) | 3 (4)
Sinus pain (Nervous system disorders) | 1 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, redness (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, erythema of right foot (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 1 (1) — small, painless pimple on testicle
Skin infection (Infections and infestations) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
White blood cell decreased (Investigations) | 2 (2)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT02153918/Prot_SAP_ICF_000.pdf